CLINICAL TRIAL: NCT06774651
Title: Comparison of Femto LDV Z8 Corneal Lenticule Extraction for Advanced Refractive Correction (CLEAR) and Visumax Small Incision Lenticule Extraction (SMILE)
Status: Recruiting | Type: Observational
Sponsor: Singapore Eye Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: R1816/58/2021
Record Dates: First submitted 2024-12-30; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Myopia
Keywords: CLEAR; FEMTO LDV Z8; SMILE; Visumax; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (2):
- 1. CLEAR surgery eyes: Eyes that have undergone CLEAR procedures.
  Interventions: Procedure: Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR)
- 2. SMILE surgery eyes: Eyes that have undergone SMILE procedures.
  Interventions: Procedure: Procedure: Small Incision Lenticule Extraction (SMILE)

INTERVENTIONS:
Procedure: Procedure: Corneal lenticule extraction for advanced refractive correction (CLEAR) — Routinely conducted procedure using FEMTO LDV Z8 laser system for correction of Myopia.
  Groups: 1. CLEAR surgery eyes
Procedure: Procedure: Small Incision Lenticule Extraction (SMILE) — Routinely conducted procedure using VisuMax laser system for correction of Myopia.
  Other Names: SMILE
  Groups: 2. SMILE surgery eyes

SUMMARY:
This observational study aims to compare two laser corrective procedures for treating myopia and myopic astigmatism: a novel refractive technique, the CLEAR procedure, and the established SMILE procedure. Participants will be randomized to undergo CLEAR in one eye and SMILE in the other. The investigators will evaluate and compare the two procedures based on the following aspects: refractive predictability (how accurate the vision correction is) by measuring the proportion of eyes close to the target prescription after surgery, clinical dry eye outcomes, changes in tear proteins, and corneal nerve changes at 1, 3, 6, and 12 months after both surgeries. Metabolomic features of the removed corneal tissue and how precisely the laser is centered during surgery will also be examined. Our hypothesis is that CLEAR provides equally good vision results as SMILE, and explore any extra benefits of CLEAR.

DETAILED DESCRIPTION:
Surgical correction for refractive errors may be performed by a number of procedures. Laser correction involves refractive procedures such as laser assisted in-situ keratomileusis (LASIK), small incision lenticule extraction (SMILE), flap based refractive lenticule extraction (femtosecond lenticule extraction and pseudo-SMILE), surface ablation techniques like photorefractive keratectomy or laser epithelial keratomileusis, while lens-based corrections involve the use of phakic intra-ocular lenses.

SMILE (Visumax) is a flapless refractive procedure which was introduced in 2011 for the treatment of myopia and myopic astigmatism. In this procedure a stromal lenticule is extracted through a small incision (2.0 to 5.0 mm). It involves docking, femtosecond laser application, lenticule dissection from the surrounding stroma, and extraction. Studies have suggested that using a SMILE technique resulted in better ocular surface stability and biomechanical strength when compared with LASIK. SMILE has a steep learning curve. The most common complication encountered during the initial learning curve, is difficult lenticule dissection and extraction with an incidence of up to 16%. Other intraoperative complications include suction loss, an opaque bubble layer, and tearing of the lenticule.

Corneal Lenticule Extraction for Advanced Refractive Correction (CLEAR) by FEMTO LDV Z8 (Ziemer) is a novel technique of flapless refractive surgery which uses low energy femtosecond laser. It creates highly focused laser pulses achieving photodisruption in the low nanojoules range (<100 nJ). Decreased stromal gas generation and accurate laser focus are the advantages of this low energy concept. The advantages of CLEAR treatment are possibility of recentering the treatment area after having performed the docking, which is not possible with the VisuMax Laser System, multiple corneal incisions for easy removal of the lenticule for the beginners, trusted vacuum with minimal suction losses. Previous study concluded that the mean preoperative sphere, cylinder, and spherical equivalents were -3.05 (D), 0.50 D, and -3.30 D respectively and 1 month after CLEAR the sphere, cylinder and spherical equivalents were 0.05 D, 0.3 D and 0.12 D respectively.

As the investigators do not expect to see a great improvement to the results from the already established SMILE procedure, the investigators aim to demonstrate that CLEAR is just as good in terms of visual outcomes. However, the investigators aim to show that CLEAR has additional benefits, on top of the equal or comparative visual outcomes.

Currently there are no publications comparing the refractive predictability, higher order aberrations, changes in tear neuromediators, tear proteomics, keratocytes and nerve regeneration, corneal lenticule metabolomics, intraoperative laser centration comparing CLEAR and SMILE, hence this study will be unique in the fact that the paired eye approach will act as an internal patient control to assess the objective and subjective outcomes in patients following both these procedures.

ELIGIBILITY:
Inclusion Criteria:

* >/= 21 years of age and </= 50 years of age.
* Cycloplegic spherical equivalent of >-1.00D
* Refractive cylinder -2.00 D or less; anisometropia <1.00D
* Best spectacle corrected visual acuity (BSCVA) of 6/12 or better in BOTH eyes.
* Spherical or cylindrical error has progressed at -0.50D or less per year from date of baseline measurement.
* Contact lens wearers must have removed contact lenses at least two (2) weeks before the baseline measurement.
* No evidence of irregular astigmatism on corneal topography.
* Available to attend post-operative examinations for a 12-month period.

Exclusion Criteria:

* Progressive or unstable myopia and/or astigmatism.
* Clinical or corneal topographic evidence of keratoconus.
* Patients who want bilateral SMILE procedure
* Patients who want extracted corneal lenticule to be stored for future refractive surgery.
* Residual, recurrent or active ocular disease such as uveitis, severe dry eyes, severe allergic eye disease, glaucoma, visually significant cataract and retinal disease.
* Previous corneal surgery or trauma within the corneal treatment zone.
* Corneal vascularisation within 1mm of the corneal treatment zone.
* Taking systemic medications likely to affect wound healing, such as corticosteroids and antimetabolites.
* Systemically immunocompromised.
* Systemic disease likely to affect wound healing, such as diabetes, connective tissue disease and severe atopy.
* Pregnant or nursing.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 65 subjects (130 eyes- 65 CLEAR eyes and 65 SMILE eyes) will be recruited in the study from refractive clinic at Singapore National Eye Centre.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of refractive predictability | 1 year
  Refractive predictability is defined as the proportion number of eyes achieving a postoperative spherical equivalent (SE) within ±1.0 D of the intended target. Uncorrected visual acuity (UCVA), refraction, and best corrected visual acuity (BCVA) will be recorded.

SECONDARY OUTCOMES:
Level of higher order aberrations | 1 year
  Higher-order aberrations are small optical irregularities of the eye that cannot be corrected with regular spectacles and most contact lenses. HOAs are responsible for an array of visual symptoms such as difficulty seeing at night, glare, halos, blurring, starburst patterns, or double vision.
Tear Break Up Time (TBUT) | 1 year
  TBUT will be measured by determining the time interval between a complete blink and the first appearance of a dry spot on the corneal surface, indicating tear film stability.
Concentration of tear neuromediators assessed by enzyme-linked immunosorbent assay | 1 year
  Tear fluid samples will be collected by the strips from Schirmer's I test. The neuromediators concentration in all tear samples will be analyzed using the enzyme-linked immunosorbent assay
Corneal sensitivity measurements assessed by Cochet-Bonnet esthesiometer | 1 year
  Corneal sensitivity measurements assess the responsiveness of the cornea to external stimuli using a contact esthesiometer (Cochet-Bonnet), evaluating the functional status of corneal nerves.
NEI score | 1 year
  Corneal fluorescein staining
Oxford grading | 1 year
  Corneal and conjunctival staining
Ocular Surface Disease Index (OSDI) questionnaire to measure eye symptoms and the impact of quality of life | 1 year
  The Ocular Surface Disease Index questionnaire is a 12-item questionnaire that used to assess the eye symptoms and and their impact on vision-related quality of life. The total Ocular Surface Disease Index score (ranging between 0 and 100) is used for evaluation, with higher scores representing greater severity of symptoms.
Extent of keratocytes activation | 1 year
  In vivo confocal microscopy will be used to capture images of keratocytes at the surgical interface, with different hyperreflective states indicating varying degrees of keratocyte activation.
Laser centration accuracy measured by the offset between the optical zone center and corneal vertex | 1 year
  Functional optical zone will be calculated using the software on Pentacam refractive power maps. Centration accuracy will be evaluated by the linear distance between the functional optical zone centroid and the corneal vertex.
Metabolites profiles of corneal lenticule | 1 year
  Metabolomic analysis technique will be used to identify and quantify small molecules in the corneal lenticule, helping to understand metabolic pathways and physiological processes related to surgeries.
Amount of tear production measured by Schirmer's I test | 1 year
  Schirmer's I test is a diagnostic method used to measure tear production by placing a standard 5 mm wide Test Strips inside the lower lid margin and assessing the amount of tear absorbed over 5 minutes.
Abundance of tear proteins assessed by quantitative proteomic analysis | 1 year
  Tear fluid samples will be collected by the strips from Schirmer's I test. Quantitative proteomic analysis technique will be used to measure and compare the abundance of proteins across different samples, providing insights into protein expression, functions, and molecular interactions.
Ocular Pain Assessment Survey (OPAS) questionnaire to measure eye pain | 1 year
  The Ocular Pain Assessment Survey (OPAS) is a 27-item questionnaire to evaluate the eye pain from 6 dimensions, including pain intensity for the last 24h, pain intensity for the last 2 weeks, non-eye pain intensity, quality of life, aggravating factors, associated factors and symptom relief. Each question was scored on a scale of 0-10, with higher score representing worse pain.
Extend of corneal nerve impairment | 1 year
  IVCM will be used to capture corneal nerve images before and after surgeries. The extend of corneal nerve damage following surgery will be quantified using seven nerve parameters by a specialized image analysis software (ACCMetrics software).

CONTACTS AND LOCATIONS:
Overall Officials: Jodhbir S Mehta, MD, FRCS, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu M, Liu C, Lee IXY, Hsu VW, Wong RKT, Anam A, Lim R, Mehta JS, Liu YC. Randomized controlled trial on corneal denervation, neuroinflammation and ocular surface in corneal lenticule extraction for advanced refractive correction (CLEAR) and small incision lenticule extraction (SMILE). Eye Vis (Lond). 2025 Apr 1;12(1):12. doi: 10.1186/s40662-025-00429-1. PMID 40165267